CLINICAL TRIAL: NCT02603419
Title: A PHASE 1 PHARMACOKINETIC-PHARMACODYNAMIC STUDY OF AVELUMAB (MSB0010718C) IN PATIENTS WITH PREVIOUSLY TREATED ADVANCED STAGE CLASSICAL HODGKIN'S LYMPHOMA
Brief Title: Avelumab In Patients With Previously Treated Advanced Stage Classical Hodgkin's Lymphoma (JAVELIN HODGKINS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to lack of recruitment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991007; 2015-002636-41 (EudraCT Number); JAVELIN HODGKINS (Other: Alias Study Number); JAVELIN HODGKIN'S (Other: Alias Study Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hodgkins Lymphoma
Keywords: classical Hodgkins Lymphoma (relapsed/refractory); post-allogeneic HSCT; anti PD-L1; Phase 1; PK; Receptor occupancy; Immunophenotypic biomarkers
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Lead-in phase-Cohort A (Experimental): X1 mg IV every 2 weeks
  Interventions: Drug: Avelumab
- Lead-in phase-Cohort B (Experimental): X2 mg IV every 2 weeks
  Interventions: Drug: Avelumab
- Lead-in phase-Cohort C (Experimental): X3 mg IV every 3 weeks
  Interventions: Drug: Avelumab
- Lead-in phase-Cohort D (Experimental): X4 mg IV every 2 weeks
  Interventions: Drug: Avelumab
- Lead-in phase-Cohort E (Experimental): X5 mg IV every 2 weeks
  Interventions: Drug: Avelumab
- Expansion phase (Experimental): X1 mg IV every 2 weeks followed by X1 or X4 mg every 2 weeks
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Anti-PD-L1 antibody at X1 mg IV every 2 weeks to optimize dosing for expansion. Treatment with avelumab will continue until disease progression.
  Arms: Lead-in phase-Cohort A
Drug: Avelumab — Anti-PD-L1 antibody at X2 mg IV every 2 weeks to optimize dosing for expansion. Treatment with avelumab will continue until disease progression.
  Arms: Lead-in phase-Cohort B
Drug: Avelumab — Anti-PD-L1 antibody at X3 mg IV every 3 weeks to optimize dosing for expansion. Treatment with avelumab will continue until disease progression
  Arms: Lead-in phase-Cohort C
Drug: Avelumab — Anti-PD-L1 antibody at X3 mg IV every 2 weeks to optimize dosing for expansion. Treatment with avelumab will continue until disease progression
  Arms: Lead-in phase-Cohort D
Drug: Avelumab — Anti-PD-L1 antibody at X mg IV every 2 weeks. Treatment with avelumab will continue until disease progression
  Arms: Lead-in phase-Cohort E
Drug: Avelumab — Anti-PD-L1 antibody at X1 mg IV every 2 weeks which can be escalated to X4 mg every 2 weeks based on safety and efficacy. Treatment with avelumab will continue until disease progression.
  Arms: Expansion phase

SUMMARY:
This is a Phase 1b, open-label, multi-center study comprising a lead-in phase and an expansion phase. The lead-in phase is a multiple-dose, randomized, parallel-arm, pharmacokinetic and pharmacodynamic study of avelumab as a single agent in adult patients with cHL. Patients enrolled in the lead-in phase of this study are required to have relapsed following a prior autologous or allogeneic HSCT, or to be ineligible for HSCT. Based on the preliminary TO, safety, and efficacy results from the lead-in phase, the expansion phase will evaluate the anti-tumor activity and safety of single-agent avelumab utilizing an intra-patient dose escalation paradigm based on two of the dosing regimens studied in the lead-in phase in 40 cHL patients in whom an allogeneic HSCT has failed.

ELIGIBILITY:
KEY INCLUSION CRITERIA

* Histological confirmation of classical Hodgkin's Lymphoma (cHL) with relapsed or refractory disease who, for the lead-in phase, either have had a prior autologous or allogeneic HSCT or are not eligible for HSCT, and , for the expansion phase, have had a prior allogeneic HSCT. In the expansion phase there must be a documented CD3+ donor chimerism of ≥20%.
* Patients must be off previous cHL therapy for at least 28 days prior to randomization in the lead-in phase/first dose of study treatment in the expansion phase.
* At least 1 fluorodeoxyglucose (FDG) PET avid (Deauville 4/5) measurable lesion >1.5 cm on PET-CT scan as defined by the Response Criteria for Malignant Lymphoma (for the lead-in phase) and the Lugano Classification (for the expansion phase) that has not previously been irradiated.
* Expansion phase: Required "de novo" or "archival" tumor biopsy, as well as required on treatment biopsy
* Estern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

KEY EXCLUSION CRITERIA

* Patients with prior allogeneic Hematopoietic Stem Cell Transplantation (allo-HSCT) who have had:

  1. Lead-in phase: allo HSCT performed <12 months prior to randomization. Expansion phase: allo-HSCT performed ≤4 months prior to the first dose of study treatment. NOTE: Patients who have had allo-HSCT performed >4 months prior to the first dose of study treatment must have discontinued all immunosuppressive therapy, and must have no clinical evidence of GVHD; or
  2. Immunosuppressive treatment for acute or chronic GVHD within 3 months prior to randomization for the lead-in phase or prior to the first dose of study treatment for the expansion phase (with the exception of those patients who required 15 mg/day oral prednisone or equivalent). Patients who required 15 mg/day oral prednisone or equivalent must have discontinued it within 7 days prior to first dose of study treatment; or
  3. Acute Grade 3 or Grade 4 GVHD at any time in the past (as defined by the modified Seattle Glucksberg criteria (Consensus Conference on Acute GVHD Grading Criteria); or
  4. Prior chronic GVHD (as defined by the NIH Consensus Development Project) that persisted for >6 months and required systemic immunosuppression (with the exception of those patients who required 15 mg/day oral prednisone or equivalent). Patients who required 15 mg/day oral prednisone or equivalent must have discontinued it within 7 days prior to the first dose of study treatment; or
  5. A donor lymphocyte infusion (DLI) within 3 months prior to randomization for the lead-in phase or first dose of study treatment for the expansion phase.
* Prior therapy with an anti PD 1 or anti PD L1 mAb.

  1. Lead-in Phase: May be enrolled if patient stopped prior anti PD1 or anti-PD-L1 therapy more than one year prior to randomization and had a documented prior response.
  2. Expansion Phase: Prior therapy with an anti-PD-1 or anti-PD-L1 agent following allo-HSCT is prohibited unless the therapy was stopped more than one year prior to the first dose of study treatment, and the patient had a documented prior response. NOTE: Prior therapy with an anti-PD-1 or anti-PD-L1 agent prior to allo-HSCT is permitted with no time limits and irrespective of a documented response.
  3. Patients with a history of ≥Grade 3 anti-PD-1 or anti-PD-L1-related immune toxicity are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- City of Hope, Duarte, California, United States
- Italy (2):
  - Az. Ospedaliera-Univers. di Bologna Policlinico S.Orsola-Malpighi, Bologna, BO
  - Istituto Clinico Humanitas U.O. Oncologia ed Ematologia, Rozzano, Milano
- United Kingdom (9):
  - Q2 Solutions, Rosebank, Livingston
  - Oxford University Hospitals NHS Foundation Trust, Headington
  - Leeds Teaching Hospital NHS Trust, Leeds
  - St James's University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - University College London Hospitals NHS Foundation Trust, London
  - UCLH Clinical Research Facility, London
  - The Christie NHS Foundation Trust, Manchester
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Herrera AF, Burton C, Radford J, Miall F, Townsend W, Santoro A, Zinzani PL, Lewis D, Fowst C, Brar S, Huang B, Thall A, Collins GP. Avelumab in relapsed/refractory classical Hodgkin lymphoma: phase 1b results from the JAVELIN Hodgkins trial. Blood Adv. 2021 Sep 14;5(17):3387-3396. doi: 10.1182/bloodadvances.2021004511. PMID 34477818
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted in 2 phases: lead-in and expansion. Expansion phase was terminated by the sponsor on 30 April 2018.
Groups:
- Lead-in Phase: Avelumab 70 mg Q2W: Participants with relapsed/refractory Classical Hodgkins Lymphoma (cHL) received an intravenous (IV) infusion of 70 milligrams (mg) of avelumab, every two weeks (Q2W) until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 47.1 weeks.
- Lead-in Phase: Avelumab 350 mg Q2W: Participants with relapsed/refractory cHL received an IV infusion of 350 mg of avelumab, Q2W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was of 123 weeks.
- Lead-in Phase: Avelumab 500 mg Q3W: Participants with relapsed/refractory cHL received an IV infusion of 500 mg of avelumab, every 3 weeks (Q3W) until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 51.1 weeks.
- Lead-in Phase: Avelumab 500 mg Q2W: Participants with relapsed/refractory cHL received an IV infusion of 500 mg of avelumab, Q2W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was of 78 weeks.
- Lead-in Phase: Avelumab 10 mg/kg Q2W: Participants with relapsed/refractory cHL received an IV infusion of 10 milligrams/kilogram (mg/kg) of avelumab, Q2W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 38.1 weeks.
- Expansion Phase: Avelumab 70 mg, 500 mg Q2W: All participants received an initial dose of 70 mg Q2W avelumab for 3 cycles, Each cycle was of 14 days (2 weeks), and were monitored for safety and efficacy. Participants who achieved a complete response (CR) at the 6-week tumor assessment were continued at the same dose regimen. Participants who achieved a partial response (PR) at 6 weeks were continued at 70 mg Q2W for an additional 3 cycles, and if the 12-week tumor assessment still showed a PR, participants were dose escalated to 500 mg Q2W. Participants who achieved a stable disease (SD) at the 6-week tumor assessment, dose escalated to 500 mg Q2W. Treatment was continued until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination the Sponsor, whichever occurred first. Maximum treatment exposure was of 48 weeks.
Period: Lead-in Phase:Maximum Exposure:123Weeks
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Started | 6 | 7 | 6 | 6 | 6 | 0
Treated | 6 | 6 | 6 | 6 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 6 | 6 | 6 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 4 | 2 | 4 | 3 | 0
Not completed — Adverse Event | 2 | 0 | 3 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0
Period: Expansion Phase:Maximum Exposure:48Weeks
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Started | 0 | 0 | 0 | 0 | 0 | 3 (Participants started expansion phase while other few participants were completing lead-in phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Lead-in Phase: Avelumab 70 mg Q2W: Participants with relapsed/refractory cHL received an IV infusion of 70 mg of avelumab, Q2W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 47.1 weeks.
- Lead-in Phase: Avelumab 500 mg Q3W: Participants with relapsed/refractory cHL received an IV infusion of 500 mg of avelumab, Q3W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 51.1 weeks.
- Lead-in Phase: Avelumab 10 mg/kg Q2W: Participants with relapsed/refractory cHL received an IV infusion of 10 mg/kg of avelumab, Q2W until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the Sponsor, whichever occurred first. Maximum treatment exposure was approximately of 38.1 weeks.
- Expansion Phase: Avelumab 70 mg, 500 mg Q2W: All participants received an initial dose of 70 mg Q2W avelumab for 3 cycles, Each cycle was of 14 days (2 weeks), and were monitored for safety and efficacy. Participants who achieved a CR at the 6-week tumor assessment were continued at the same dose regimen. Participants who achieved a PR at 6 weeks were continued at 70 mg Q2W for an additional 3 cycles, and if the 12-week tumor assessment still showed a PR, participants were dose escalated to 500 mg Q2W. Participants who achieved a SD at the 6-week tumor assessment, dose escalated to 500 mg Q2W. Treatment was continued until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination the Sponsor, whichever occurred first. Maximum treatment exposure was of 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W | Expansion Phase: Avelumab 70 mg, 500 mg Q2W | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 3 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 6 | 5 | 3 | 28
  >=65 years | 1 | 2 | 2 | 0 | 1 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 1 | 2 | 9
  Male | 3 | 6 | 5 | 5 | 5 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 7 | 5 | 6 | 5 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 0 | 0 | 0 | 0 | 3
  White | 4 | 5 | 5 | 4 | 5 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Lead-in Phase: Percent Target Occupancy (CD14+ Monocytes) at Day 2 of Cycle 1
Description: Target occupancy on peripheral blood CD14+ T-cells by avelumab was investigated in human blood in vitro by flow cytometry.
Time Frame: Day 2 of Cycle 1
Population: The Target Occupancy (TO) analysis set included all participants who received at least one dose of study drug and who had at least one receptor occupancy blood sample collected both pre and post Cycle 1 Day 1 dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of occupancy
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 5
percentage of occupancy | 99.5 (0.01) | 97.7 (0.02) | 97.6 (0.03) | 99.7 (0.00) | 97.8 (0.03)

2. Primary Outcome: Lead-in Phase: Percent Target Occupancy (CD14+ Monocytes) at Day 1 of Cycle 2
Description: as for outcome 1
Time Frame: Day 1 of Cycle 2
Population: The TO analysis set included all participants who received at least one dose of study drug and who had at least one receptor occupancy blood sample collected both pre and post Cycle 1 Day 1 dose. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of occupancy
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 4 | 6 | 4 | 4 | 4
percentage of occupancy | 96.3 (0.04) | 96.2 (0.08) | 97.0 (0.04) | 97.3 (0.05) | 98.8 (0.02)

3. Primary Outcome: Lead-in Phase: Percent Target Occupancy (CD3+ T-Cells) at Day 2 of Cycle 1
Description: Target occupancy on peripheral blood CD3+ T-cells by avelumab was investigated in human blood in vitro by flow cytometry.
Time Frame: Day 2 of Cycle 1
Population: The TO analysis set included all participants who received at least one dose of study drug and who had at least one receptor occupancy blood sample collected both pre and post Cycle 1 Day 1 dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of occupancy
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 5
percentage of occupancy | 99.0 (0.01) | 99.0 (0.02) | 96.8 (0.05) | 99.7 (0.01) | 89.8 (0.22)

4. Primary Outcome: Lead-in Phase: Percent Target Occupancy (CD3+ T-Cells) at Day 1 of Cycle 2
Description: as for outcome 3
Time Frame: Day 1 of Cycle 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of occupancy
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 4 | 6 | 4 | 4 | 4
percentage of occupancy | 81.7 (0.37) | 91.9 (0.14) | 99.1 (0.02) | 99.7 (0.01) | 98.7 (0.01)

5. Primary Outcome: Expansion Phase: Percentage of Participants With Objective Response as Assessed by Blinded Independent Central Review (BICR)
Description: Objective response: complete response (CR) or partial response (PR) according to the Response Criteria for Malignant Lymphoma, from 'start date' until disease progression (Disease progression: >= 20% and >= 5-mm increase in sum of target lesion diameters in reference to smallest sum on study and/or substantial worsening in non-target disease) or death due to any cause. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in sum of products of greatest diameters. PR was defined >= 50% decreased in the sum of products of the greatest diameters (SPD) of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.
Time Frame: From treatment start in expansion phase until progressive disease or death due to any cause (maximum duration of 14 months)
Population: Data for this outcome measure (OM) was not collected due to the limited number of participants were enrolled into the expansion phase prior to study termination.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

6. Primary Outcome: Lead-in Phase: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinity (AUC0-inf) of Avelumab After Single Dose
Description: AUC(0-inf) was defined as area under the plasma concentration-time profile from time zero to extrapolated infinity AUC(0-inf), after single dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 1
Population: The PK parameter analysis set included all participants who received at least one dose of study drug and those who had at least one of the PK parameters of interest for avelumab. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/mL (hr*mcg/mL)
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 5
hour*microgram/mL (hr*mcg/mL) | 2588 (59) | 8600 (40) | 15887 (29) | 17647 (55) | 23789 (61)

7. Primary Outcome: Lead-in Phase: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinity (AUC0-inf) of Avelumab After Multiple Dose
Description: AUC(0-inf) was defined as area under the plasma concentration-time profile from time zero to extrapolated infinity AUC(0-inf), after multiple dose.
Time Frame: pre-dose, 1, 6, 24, 144, 312, 336 and 504 hours post-dose on Day 1 of Cycle 2
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Lead-in Phase: Maximum Observed Plasma Concentration (Cmax) of Avelumab After Single Dose
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 3
micrograms per milliliter (mcg/mL) | 24.0 (35) | 68.4 (33) | 126 (15) | 143 (24) | 271 (16)

9. Primary Outcome: Lead-in Phase: Maximum Observed Plasma Concentration (Cmax) of Avelumab After Multiple Dose
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2
mcg/mL | 26.1 (21) | 78.7 (19) | 135 (8) | 195 (46) | 273 (22)

10. Primary Outcome: Lead-in Phase: Area Under the Plasma Concentration-Time Profile From Time Zero (Pre-Dose) to the Next Dose (AUC0-tau) of Avelumab After Single Dose
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero (pre-dose) to the next dose (AUC0-tau) of avelumab, after single dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6
hr*mcg/mL | 1933 (64) | 8450 (28) | 15392 (27) | 15436 (38) | 23780 (54)

11. Primary Outcome: Lead-in Phase: Area Under the Plasma Concentration-Time Profile From Time Zero (Pre-Dose) to the Next Dose (AUC0-tau) of Avelumab After Multiple Dose
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero (pre-dose) to the next dose (AUC0-tau) of avelumab, after multiple dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 5
hr*mcg/mL | 2067 (6) | 8789 (39) | 19173 (23) | 21053 (47) | 27196 (59)

12. Primary Outcome: Lead-in Phase: Terminal Elimination Half-Life (t1/2) of Avelumab After Single Dose
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half of avelumab, after single dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 4 | 6 | 5 | 5
days | 3.49 (28) | 3.25 (44) | 4.04 (23) | 4.38 (39) | 3.88 (38)

13. Primary Outcome: Lead-in Phase: Terminal Elimination Half-Life (t1/2) of Avelumab After Multiple Dose
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half of avelumab, after multiple dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 5
days | 2.92 (13) | 3.43 (43) | 4.62 (17) | 4.59 (36) | 4.23 (37)

14. Primary Outcome: Lead-in Phase: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Avelumab After Single Dose
Description: Time to reach maximum observed plasma concentration of avelumab, after single dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 3
hours | 1.13 [1.00 to 1.22] | 21.60 [5.78 to 25.10] | 1.99 [1.23 to 24.30] | 1.59 [1.17 to 2.00] | 1.50 [1.17 to 6.08]

15. Primary Outcome: Lead-in Phase: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Avelumab After Multiple Dose
Description: Time to reach maximum observed plasma concentration of avelumab, after multiple dose.
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2
hours | 1.18 [1.02 to 2.00] | 1.48 [0.97 to 7.00] | 1.32 [1.17 to 2.00] | 1.53 [0.98 to 2.00] | 6.71 [6.67 to 6.75]

16. Primary Outcome: Lead-in Phase: Pre-Dose Concentration During Multiple Dosing (Ctrough) of Avelumab After Multiple Dose
Time Frame: pre-dose, 1, 6, 24, 144, and 312 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 4 | 6 | 5 | 6 | 6
mcg/mL | 1.71 (163) | 4.03 (110) | 2.54 (125) | 12.1 (93) | 14.4 (170)

17. Primary Outcome: Lead-in Phase: The Last Time Point of the Last Quantifiable Concentration (Tlast) of Avelumab After Single Dose
Description: The last time point of the last quantifiable concentration (Tlast) of avelumab, after single dose.
Time Frame: pre-dose, 1, 6, 24, 144, 312 and 527 hours post-dose on Day 1 of Cycle 1
Population: The PK parameter analysis set included all participants who received at least one dose of study drug and those who had at least one of the PK parameters of interest for avelumab.
Measure: Median (Full Range); unit: hours
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
hours | 168.00 [26.50 to 336.00] | 335.00 [165.00 to 336.00] | 504.50 [312.00 to 527.00] | 334.50 [333.00 to 357.00] | 335.50 [290.00 to 360.00]

18. Primary Outcome: Lead-in Phase: The Last Time Point of the Last Quantifiable Concentration (Tlast) of Avelumab After Multiple Dose
Description: The last time point of the last quantifiable concentration (tlast) of avelumab, after multiple dose.
Time Frame: pre-dose, 1, 6, 24, 144, 312, 336 and 504 hours post-dose on Day 1 of Cycle 2
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Lead-in Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Related TEAEs and TEAEs Graded >=3 as Per National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03: Grade 3: severe or medically significant but not immediately life-threatening, or prolongation of existing hospitalization indicated; Grade 4: life-threatening consequence; Grade 5: death related to AE. SAE was an AE resulting in any of following outcomes: death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or congenital anomaly. A TEAEs: an event that emerged during treatment period (From first dose of study drug until end of open label phase [From first dose of study drug to 90 days after last administration of study drug (maximum duration of 32 months)] that was absent before treatment,or worsened during treatment period relative to pre-treatment state. AE was considered related to study drug if event was assessed by investigator as probably or possibly related.
Time Frame: From first dose of study drug to 90 days after last administration of study drug (maximum duration of 32 months)
Population: Safety analysis set included all participants who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants
  AEs | 6 | 6 | 6 | 6 | 6
  SAEs | 5 | 2 | 3 | 2 | 0
  Related TEAEs | 6 | 6 | 6 | 4 | 4
  TEAEs Graded >=3 | 6 | 3 | 2 | 5 | 1

20. Secondary Outcome: Lead-in Phase: Number of Participants With Laboratory Abnormalities Graded Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: Hematology: Anemia (Grade)G3: Hg <8.0 grams/deciliter (g/dL); lymphocyte count decreased G3: <0.5-0.2*10^9/L, G4: <0.2*10^9/L; neutrophil count decreased: G3: <1.0-0.5*10^9/L, G4: <0.5*10^9/L; platelet count decreased: G3:<50.0-25.0*10^9/L, G4: <25.0*10^9/L; white blood cell (WBC) decreased: G3: <0.2*10^9/L, G4: <1.0*10^9/L. Chemistry: [ALT, ALP increased and AST G3: >5.0-20.0*ULN, G4: >20.0*ULN]. blood bilirubin increased: G3: >3.0-10.0*ULN, G4: >10.0 *ULN. [cholesterol high: G3: >10.34 - 12.92, G4: >12.92; hypokalemia G3: <3.0-2.5, G4: <2.5]mmol/L, creatine phosphokinase (Cpk) increased: G3: >5*ULN-10*ULN, G4: >10*ULN; gamma-glutamyl transferase (Ggt) increased: G3: >5.0-20.0*ULN, G4: >20.0*ULN; [hypertriglyceridemia G3: >500-1000, G4: >1000; hypermagnesemia, G3: >3.0-8.0, G 4: >8.0]mg/dL, Lipase increased: G3: >2.0 - 5.0*ULN, G4: >5.0*ULN, Serum amylase increased: G3: >2.0 - 5.0*ULN, G4: >5.0*ULN. Only those category in which at least one participant had data were reported.
Time Frame: From first dose of study drug up to 90 days after the last administration of the study drug (maximum duration of 32 months)
Population: Safety analysis set included all participants who receive at least one dose of study drug. Here, 'Number analyzed' ('n') = Participants evaluable for this outcome measure for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants
  Anemia | 0 | 1 | 0 | 0 | 0
  Lymphocyte count decreased | 2 | 0 | 0 | 1 | 1
  Neutrophil count decreased | 1 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 1 | 2 | 1 | 0
  White blood cell decreased | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase (ALT)increased: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Alanine aminotransferase (ALT)increased | 2 | 0 | 0 | 1 | 0
  Alkaline phosphatase (ALP) increased: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Alkaline phosphatase (ALP) increased | 2 | 1 | 1 | 0 | 0
  Aspartate aminotransferase (AST) increased: number analyzed (Participants) | 4 | 6 | 6 | 5 | 5
  Aspartate aminotransferase (AST) increased | 2 | 0 | 0 | 0 | 0
  Blood bilirubin increased: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Blood bilirubin increased | 1 | 0 | 1 | 0 | 0
  Cholesterol high: number analyzed (Participants) | 4 | 6 | 5 | 5 | 5
  Cholesterol high | 1 | 0 | 0 | 0 | 0
  Cpk increased: number analyzed (Participants) | 4 | 6 | 6 | 6 | 6
  Cpk increased | 0 | 1 | 0 | 0 | 0
  Ggt increased: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Ggt increased | 2 | 1 | 2 | 0 | 0
  Hypermagnesemia: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Hypermagnesemia | 0 | 1 | 0 | 0 | 0
  Hypertriglyceridemia: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Hypertriglyceridemia | 0 | 1 | 1 | 0 | 0
  Hypokalemia: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Hypokalemia | 0 | 0 | 1 | 0 | 0
  Lipase increased: number analyzed (Participants) | 4 | 6 | 5 | 5 | 6
  Lipase increased | 1 | 0 | 1 | 1 | 0
  Serum amylase increased: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Serum amylase increased | 1 | 0 | 0 | 0 | 0

21. Secondary Outcome: Lead-in Phase: Number of Participants With Anti-Drug Antibodies (ADA) Status
Description: ADA against avelumab in serum samples was determined and reported separately for ADA never-positive and ADA ever-positive participants. ADA never-positive participants were those who had no positive (titer less than cutpoint [22.5 percentage (%) inhibition]) ADA results at any time point. ADA ever-positive participants were defined as those who had at least one positive (titer greater than or equal to cutpoint [22.5% inhibition]) ADA result at any time point.
Time Frame: Day 1 up to Month 29
Population: The immunogenicity analysis set included all participants who received at least one dose of study drug and who had at least one ADA sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
Participants
  ADA never-positive | 5 | 5 | 3 | 4 | 6
  ADA ever-positive | 0 | 1 | 3 | 2 | 0

22. Secondary Outcome: Expansion Phase: Number of Participants With Anti-Drug Antibodies (ADA) Status
Description: ADA against avelumab in serum samples was determined and reported separately for ADA never-positive and ADA ever-positive participants. ADA never-positive participants were those who had no positive (titer less than cutpoint [22.5% inhibition]) ADA results at any time point. ADA ever-positive participants were defined as those who had at least one positive (titer greater than or equal to cutpoint [22.5% inhibition]) ADA result at any time point.
Time Frame: Day 1 up to Month 14
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 3
Participants
  ADA never-positive | 2
  ADA ever-positive | 1

23. Secondary Outcome: Lead-in Phase: Number of Participants With Neutralizing Antibodies (nAb) Status
Description: nAb against avelumab in serum samples was determined and reported separately for nAb never-positive and nAb ever-positive participants. nAb never-positive participants were those who had no positive (titer less than cutpoint [0.71]) nAb results at any time point. nAb ever-positive participants were defined as those who had at least one positive (titer greater than or equal to cutpoint [0.71]) nAb result at any time point.
Time Frame: Day 1 up to Month 29
Population: The immunogenicity analysis set included all participants who received at least one dose of study drug and who had at least one nAb sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
Participants
  nAb never-positive | 5 | 5 | 4 | 6 | 6
  nAb ever-positive | 0 | 1 | 2 | 0 | 0

24. Secondary Outcome: Expansion Phase: Number of Participants With Neutralizing Antibodies (nAb) Status
Description: as for outcome 23
Time Frame: Day 1 up to Month 14
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 3
Participants
  nAb never-positive | 3
  nAb ever-positive | 0

25. Secondary Outcome: Lead-in Phase: Number of ADA Ever Positive Participants For Each Serum ADA Titers for Avelumab
Description: Serum samples were assayed for ADA using a validated analytical method. Number of ADA ever positive participants for each serum ADA titer (180, 4860, 43740 and 131220) are reported.
Time Frame: Day 1 up to Month 29
Population: Analysis was performed on participants who had received at least one dose of study drug and who had ADA ever-positive results. Here "0" in overall number of participants analyzed signifies that there were no ADA ever-positive participants in that specified group".
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 1 | 3 | 2 | 0
Participants
  180 |  | 0 | 1 | 1 |
  4860 |  | 0 | 1 | 0 |
  43740 |  | 0 | 1 | 1 |
  131220 |  | 1 | 0 | 0 |

26. Secondary Outcome: Expansion Phase: Number of ADA Ever Positive Participants For Each Serum ADA Titers for Avelumab
Description: as for outcome 25
Time Frame: Day 1 up to Month 14
Population: Analysis was performed on participants who had received at least one dose of study drug and who had ADA ever-positive results.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 1
Participants
  180 | 1
  4860 | 0
  43740 | 0
  131220 | 0

27. Secondary Outcome: Lead-in Phase: Number of nAb Ever Positive Participants For Serum nAb Titer for Avelumab
Description: Serum samples were assayed for nAb using a validated analytical method. Number of nAb ever positive participants for serum nAb titer (1) is reported.
Time Frame: Day 1 up to Month 29
Population: Analysis was performed on participants who had received at least one dose of study drug and who had nAb ever-positive results. Here "0" in overall number of participants analyzed signifies that there were no nAb ever-positive participants in that specified group.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 1 | 2 | 0 | 0
Participants | 0 | 1 | 2 | 0 | 0

28. Secondary Outcome: Expansion Phase: Number of nAb Ever Positive Participants For Serum nAb Titer for Avelumab
Description: Serum samples were assayed for nAb using a validated analytical method.
Time Frame: Day 1 up to Month 14
Population: Analysis was performed on participants who had received at least one dose of study drug and who had nAb ever-positive results. Here "0" in overall number of participants analyzed signifies that there were no nAb ever-positive participants in the specified group.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

29. Secondary Outcome: Lead-in Phase: Number of Participants With Phenotype of Tumor Infiltrating Lymphocytes (TILs) in Tumor Biopsy
Time Frame: Day 1 (pre-dose) and Day 14 of Cycle 1, Day 7 of Cycle 2, Day 1 (pre-dose) of Cycle 3, 5, 7; and at End of Treatment (EOT) (maximum duration of 29 months)
Population: Data for this outcome measure was not collected and analyzed due to lack of availability of tumor biopsy tissue for analysis.
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Lead-in Phase: Number of Participants With Gene Expression of Transcripts Associated With Immune Activation and Regulation
Time Frame: Day 1 (pre-dose) and Day 14 of Cycle 1, Day 7 of Cycle 2, Day 1 (pre-dose) of Cycle 3, 5, 7; and at End of Treatment (maximum duration of 29 months)
Population: as for outcome 29
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Lead-in Phase: Number of Participants With T Cell Immunophenotype
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 7, 10 and at End of Treatment (maximum duration of 29 months)
Population: Data for this outcome measure was not collected and analyzed, as the assay (which was planned for this parameter) could not be used due to quality issues.
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Lead-in Phase: Percentage of Participants With Objective Response as Assessed by Investigator
Description: Objective response: complete response (CR) or partial response (PR) according to the Response Criteria for Malignant Lymphoma, from 'start date' until disease progression (Disease progression: >= 20% and >= 5-mm increase in sum of target lesion diameters in reference to smallest sum on study and/or substantial worsening in non-target disease) or death due to any cause. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in sum of products of greatest diameters. PR was defined >= 50% decreased in the SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.
Time Frame: From randomization until disease progression or death due to any cause (maximum duration of 32 months)
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
percentage of participants | 33.3 [4.3 to 77.7] | 0 [0.0 to 41.0] | 83.3 [35.9 to 99.6] | 33.3 [4.3 to 77.7] | 66.7 [22.3 to 95.7]

33. Secondary Outcome: Lead-in Phase: Percentage of Participants With Disease Control (DC) as Assessed by Investigator
Description: DC: best overall response of CR, PR, or stable disease (SD). CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75% in sum of the products of greatest diameters. PR was defined >=50% decreased in SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in SPD and SD was defined as < PR but not progressive disease. To qualify as a best overall response of SD, at least one SD assessment must be observed >=6 weeks after start date and before disease progression. (Disease progression: >= 20% and >= 5-mm increase in sum of target lesion diameters in reference to smallest sum on study and/or substantial worsening in non-target disease).
Time Frame: From randomization to PD, death or start of new anti-cancer therapy (maximum duration of 32 months)
Population: FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
percentage of participants | 50.0 [11.8 to 88.2] | 57.1 [18.4 to 90.1] | 100.0 [54.1 to 100.0] | 66.7 [22.3 to 95.7] | 66.7 [22.3 to 95.7]

34. Secondary Outcome: Lead-in Phase: Time to Tumor Response (TTR) as Assessed by Investigator
Description: TTR was defined, for participants with an objective response as the time from 'start date' to the first documentation of objective tumor response (CR or PR). CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.
Time Frame: From the date of randomization to the first documentation of objective response (CR or PR) (maximum duration of 32 months)
Population: The FAS included all randomized participants. Here, Overall Number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 2 | 0 | 5 | 2 | 4
months | 2.6 [1.7 to 3.5] |  | 1.5 [1.4 to 1.6] | 1.5 [1.4 to 1.5] | 2.1 [1.4 to 2.8]

35. Secondary Outcome: Lead-in Phase: Duration of Response (DR) as Assessed by Investigator
Description: DR is defined, for participants with an objective response, as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective PD or to death due to any cause, whichever occurs first. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.(PD: >= 20% and >= 5-mm increase in sum of target lesion diameters in reference to smallest sum on study and/or substantial worsening in non-target disease).
Time Frame: From first documentation of objective response to date of first documentation of objective PD or death due to any cause (maximum duration of 32 months)
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 2 | 0 | 5 | 2 | 4
months | NA [NA to NA] — Median, upper and lower limits of 95% CI was not estimable due to smaller number of participants with the event. |  | 6.9 [4.3 to NA] — Upper limits of 95% CI was not estimable due to smaller number of participants with the event. | 6.9 [1.4 to 12.4] | 9.4 [1.8 to 9.4]

36. Secondary Outcome: Lead-in Phase: Progression-Free Survival (PFS) as Assessed by Investigator
Description: PFS was defined as time (in months) from date of randomization to the first documentation of disease progression or death (due to any cause), whichever occurred first. Progression as per RECIST 1.1, was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered as progression of disease.
Time Frame: From randomization to the date of progression of disease or death due to any cause, whichever occurs first (maximum duration of 32 months)
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
months | NA [1.7 to NA] — Median and upper limits of 95% CI was not estimable due to smaller number of participants with the event. | 5.7 [2.8 to NA] — Upper limit of 95% CI was not estimable due to smaller number of participants with the event. | 8.5 [8.5 to NA] — Upper limit of 95% CI was not estimable due to smaller number of participants with the event. | 3.1 [1.4 to 5.5] | 6.1 [1.4 to 10.8]

37. Secondary Outcome: Expansion Phase: Percentage of Participants With Objective Response as Assessed by Investigator
Description: Objective response was defined as CR or PR according to the Response Criteria for Malignant Lymphoma, from 'start date' until disease progression or death due to any cause. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the SPD of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD. (PD: >= 20% and >= 5-mm increase in sum of target lesion diameters in reference to smallest sum on study and/or substantial worsening in non-target disease).
Time Frame: From treatment start in expansion phase until disease progression or death due to any cause (maximum duration of 14 months)
Population: Data for this outcome measure was not collected due to the limited number of participants were enrolled into the expansion phase prior to study termination.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

38. Secondary Outcome: Expansion Phase: Time to Tumor Response (TTR) as Assessed by Investigator and by Blinded Independent Central Review (BICR)
Description: Time to Tumor Response (TTR) was defined, for participants with an objective response as the time from 'start date' to the first documentation of objective tumor response (CR or PR). CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the sum of products of the greatest diameters (SPD) of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.
Time Frame: From treatment start in expansion phase to first documentation of objective response (CR or PR) (maximum duration of 14 months)
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

39. Secondary Outcome: Expansion Phase: Duration of Response (DR) as Assessed by Investigator and by Blinded Independent Central Review (BICR)
Description: Duration of Response (DR) is defined, for participants with an objective response, as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective progression of disease (PD) or to death due to any cause, whichever occurs first. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the sum of products of the greatest diameters (SPD) of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD.
Time Frame: From first documentation of objective response in expansion phase to date of first documentation of objective PD or death due to any cause (maximum duration of 14 months)
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

40. Secondary Outcome: Expansion Phase: Percentage of Participants With Disease Control (DC) as Assessed by Investigator and by Blinded Independent Central Review (BICR)
Description: Disease Control (DC) was defined as the best overall response of CR, PR, or SD. CR was defined as all lymph nodes must have regressed to normal size(less than or equal to 1.5 cm in greatest diameter if >1.5 cm before therapy). Previously involved nodes that were 1.1 to 1.5 cm in greatest diameter must have decreased to less than or equal to 1 cm or by more than 75 percent in the sum of the products of the greatest diameters. PR was defined >=50% decreased in the sum of products of the greatest diameters (SPD) of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease. Splenic and hepatic nodules must regress by >=50% in the SPD and Stable Disease was defined as less than a PR but not progressive disease. To qualify as a best overall response of SD, at least one SD assessment must be observed >=6 weeks after start date and before disease progression.
Time Frame: From treatment start in expansion phase to PD, death or start of new anti-cancer therapy (maximum duration of 14 months)
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

41. Secondary Outcome: Expansion Phase: Progression-Free Survival (PFS) as Assessed by Investigator and by Blinded Independent Central Review (BICR)
Description: PFS was defined as time (in months) from date of randomization to the first documentation of disease progression or death (due to any cause), whichever occurred first. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Analysis was performed using a Cox's Proportional Hazard model stratified by the randomization strata and a stratified log-rank test.
Time Frame: From treatment start in expansion phase to date of first documentation of objective Progressive Disease (PD) or death due to any cause, whichever occurs first (maximum duration of 14 months)
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

42. Secondary Outcome: Expansion Phase: Overall Survival
Description: Overall survival was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From treatment start in expansion phase until death (maximum duration of 14 months)
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

43. Secondary Outcome: Expansion Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Related TEAEs and TEAEs Graded >=3 Based on, National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03: Grade 3: severe or medically significant but not immediately life-threatening, or prolongation of existing hospitalization indicated; Grade 4: life-threatening consequence; Grade 5: death related to AE. SAE was an AE resulting in any of following outcomes: death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or congenital anomaly. TEAEs: an event that emerged during treatment period (From first dose of study drug until end of expansion phase [From first dose of study drug to 90 days after last administration of study drug (maximum duration of 14 months)] that was absent before treatment, or worsened during treatment period relative to pre-treatment state. AE was considered related to study drug if event was assessed by investigator as probably or possibly related.
Time Frame: From first dose of study drug to 90 days after last administration of study drug (maximum duration of 14 months)
Population: Safety analysis set included all participants who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 3
Participants
  AEs | 2
  SAEs | 2
  Related TEAEs | 0
  TEAEs Graded | 0

44. Secondary Outcome: Expansion Phase: Number of Participants With Laboratory Abnormalities of Grade 3 Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: As per NCI-CTCAE v 4.03, Grade >= 3 criteria were; Alanine aminotransferase: 0 LLN, 0.58 ULN microkat/L (microkatal /L); GGT: 0 LLN, 0.63 ULN microkat/L, Glucose: 4.11 LLN, 5.88 ULN mmol/L, LOW Sodium: 136 LLN, 146 ULN mmol/L; Prothrombin intl. normalized ratio: 0.9 LLN, 1.2 ULN; LOW lymphocytes (10^9/L); 1.5 LLN, 4.0 ULN; Platelets (10^9/L): 130 LLN, 400 ULN. Only those category in which at least one participant had data were reported.
Time Frame: From first dose of study drug to 90 days after last administration of study drug (maximum duration of 14 months)
Population: Safety analysis set included all participants who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 3
Participants
  Alanine Aminotransferase | 1
  Gamma Glutamyl Transferase | 1
  Glucose | 1
  Low Sodium | 1
  Prothrombin Intl. Normalized Ratio | 1
  Platelets | 1

45. Secondary Outcome: Expansion Phase: Number of Participants With Acute and Chronic Graft Versus Host Disease (GVHD)
Description: Acute GvHD is a reaction of donor immune cells against host tissues. The three main tissues that acute GvHD affects are the skin, liver and gastrointestinal tract. Chronic GvHD is a syndrome of variable clinical features resembling autoimmune and other immunologic disorders. Manifestations of chronic GvHD may be restricted to a single organ or site or may be widespread, with profound impact on quality of life.
Time Frame: From treatment start in expansion phase up to 90 days after last administration of study drug (maximum duration of 14 months)
Population: FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 3
Participants | 0

46. Secondary Outcome: Expansion Phase: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinity (AUC0-inf), After Single and Multiple Dose
Description: AUC(0-inf) was defined as area under the plasma concentration-time profile from time zero to infinity AUC(0-inf), after single and multiple dose.
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

47. Secondary Outcome: Expansion Phase: Maximum Observed Plasma Concentration (Cmax) of Avelumab After Single and Multiple Dose
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

48. Secondary Outcome: Expansion Phase: Area Under the Plasma Concentration-Time Profile From Time Zero (Pre-Dose) to the Next Dose (AUC0-tau) of Avelumab, After Single and Multiple Dose
Description: AUCtau was defined as area under the plasma concentration-time profile from time zero (pre-dose) to the next dose (AUC0-tau) of avelumab, after single and multiple dose.
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

49. Secondary Outcome: Expansion Phase: Terminal Elimination Half-Life (t1/2) of Avelumab After Single and Multiple Dose
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

50. Secondary Outcome: Expansion Phase: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Avelumab After Single and Multiple Dose
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

51. Secondary Outcome: Expansion Phase: Pre-Dose Concentration During Multiple Dosing (Ctrough) of Avelumab After Single and Multiple Dose
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

52. Secondary Outcome: Expansion Phase: The Last Time Point of the Last Quantifiable Concentration (Tlast) of Avelumab After Single and Multiple Dose
Description: The last time point of the last quantifiable concentration (tlast), after single and multiple dose.
Time Frame: pre-dose and 1 hour post-dose on Day 1 of Cycles 1, 2 and 3
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

53. Secondary Outcome: Expansion Phase: Number of Participants With Phenotype of Tumor Infiltrating Lymphocytes (TILs) in Tumor Biopsy
Time Frame: Pre-treatment tumor biopsy for baseline and on-treatment biopsy at Day 7 of Cycle 3
Population: as for outcome 37
Arm/Group | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Lead-in phase: From first dose of study drug to 90 days after last administration of study drug (maximum duration of 32 months), Expansion phase: From first dose of study drug in expansion phase to 90 days after last administration of study drug (maximum duration of 14 months).
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non serious in another participant or 1 participant may have experienced both serious and non serious event during study.
Arm/Group | Lead-in Phase: Avelumab 70 mg Q2W | Lead-in Phase: Avelumab 350 mg Q2W | Lead-in Phase: Avelumab 500 mg Q3W | Lead-in Phase: Avelumab 500 mg Q2W | Lead-in Phase: Avelumab 10 mg/kg Q2W | Expansion Phase: Avelumab 70 mg, 500 mg Q2W
All-Cause Mortality (participants affected / at risk) | 1/6 | 4/6 | 1/6 | 4/6 | 3/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/6 | 3/6 | 2/6 | 0/6 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Phase: Avelumab 70 mg Q2W (N=6) | Lead-in Phase: Avelumab 350 mg Q2W (N=6) | Lead-in Phase: Avelumab 500 mg Q3W (N=6) | Lead-in Phase: Avelumab 500 mg Q2W (N=6) | Lead-in Phase: Avelumab 10 mg/kg Q2W (N=6) | Expansion Phase: Avelumab 70 mg, 500 mg Q2W (N=3)
Lung infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Graft versus host disease in liver (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead-in Phase: Avelumab 70 mg Q2W (N=6) | Lead-in Phase: Avelumab 350 mg Q2W (N=6) | Lead-in Phase: Avelumab 500 mg Q3W (N=6) | Lead-in Phase: Avelumab 500 mg Q2W (N=6) | Lead-in Phase: Avelumab 10 mg/kg Q2W (N=6) | Expansion Phase: Avelumab 70 mg, 500 mg Q2W (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lip exfoliation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 1 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 2 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2 | 1 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Blood viscosity increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Results for PK parameters(AUC0-inf and Tlast after Multiple Dose) in Lead-in phase and (AUC0-inf, Cmax,AUC0-tau, t1/2, Tmax, Ctrough and Tlast after single and multiple doses) in expansion phase not reported, as data for these OMs were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT02603419/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02603419/SAP_001.pdf